CLINICAL TRIAL: NCT02972671
Title: Multicenter Randomized Study of the MiStent Sirolimus Eluting Absorbable Polymer Stent System (MT005) for Revascularization of Coronary Arteries
Brief Title: Trial of MiStent Compared to Xience in Japan
Acronym: DESSOLVEJ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Micell Technologies (Industry)
Collaborators: Cardialysis BV (Industry); ClinLogix. LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MIS-JPN-2016-05
Record Dates: First submitted 2016-11-16; First posted 2016-11-23 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Coronary (Artery); Disease
Keywords: MiStent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MiStent (MT005) Coronary Artery Stent (Experimental): A balloon expandable crystalline sirolimus eluting stent with an absorbable polymer coating will be implanted.
  Interventions: Device: MiStent (MT005) Coronary Artery Stent
- Xience Coronary Artery Stent (Active Comparator): Balloon expandable drug eluting stents using everolimus with a non-erodible or durable polymer coating will be implanted
  Interventions: Device: Xience Coronary Artery Stent

INTERVENTIONS:
Device: MiStent (MT005) Coronary Artery Stent — Implantation of a coronary artery stent in an all-comers population, including patients with symptomatic coronary artery disease including patients with chronic stable angina, silent ischemia, and acute coronary syndromes, who qualify for percutaneous coronary interventions
  Arms: MiStent (MT005) Coronary Artery Stent
Device: Xience Coronary Artery Stent — Implantation of a coronary artery stent in an all-comers population, including patients with symptomatic coronary artery disease including patients with chronic stable angina, silent ischemia, and acute coronary syndromes, who qualify for percutaneous coronary interventions
  Arms: Xience Coronary Artery Stent

SUMMARY:
To compare the MT005 (MiStent) with the XIENCE with respect to target lesion failure (TLF) at 12 months in a non-inferiority trial in a "real world" patient population and to confirm that the domestic extrapolation of the DESSOLVE III study results is valid.

DETAILED DESCRIPTION:
This is a prospective, randomized, 1:1 balanced, controlled, double-blind, multi-center study comparing clinical outcomes at 12 months between MT005 (MiStent) and XIENCE in an all-comers population, including patients with symptomatic coronary artery disease including patients with chronic stable angina, silent ischemia, and acute coronary syndromes, who qualify for percutaneous coronary interventions.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥20 years;
* Patients who are eligible for percutaneous coronary intervention (PCI);
* The vessel should have a reference vessel diameter ranging from 2.5 mm to 3.75 mm. All lesions of the patient must comply with the angiographic inclusion criteria and no more than 4 stents per patient are to be implanted.
* The patient is judged to be capable of providing voluntary informed consent and has been fully informed of the nature of the study, is willing to comply with all study requirements and will provide written informed consent as approved by the Ethics Committee of the respective clinical site.

Exclusion Criteria:

* Known pregnancy or breastfeeding at time of randomization or planned pregnancy for 12 months after the index treatment. Women of childbearing potential must have a negative pregnancy test within 7 days of randomization;
* Known contraindication or hypersensitivity to sirolimus, everolimus, cobalt-chromium, or to medications such as aspirin, heparin, bivalirudin, and all of the following three medications: clopidogrel bisulfate, ticlopidine, prasugrel;
* Concurrent medical condition with a life expectancy of less than 12 months;
* The patient is unwilling/not able to return for outpatient clinic at 1, 6 and 12 months follow-up;
* Currently participating in another trial and not yet at its primary endpoint;

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF)-Composite of Target Lesion Revascularization (TLR), Target Vessel MI (TV MI), and Cardiac Death | 12 Months
  The proportion of patients in each arm that experience TLF will be summarized and reported. No formal comparison of the two arms will be conducted. Portions will be reported at 12 months post procedure.

SECONDARY OUTCOMES:
Target Lesion Revascularization (TLR) | 12 Months
  The proportion of patients in each arm that experience TLR will be summarized and reported. No formal comparison of the two arms will be conducted. Portions will be reported at 12 months post procedure.
Target Vessel Myocardial Infarction (TV-MI) | 12 Months
  The proportion of patients in each arm that experience TV-MI will be summarized and reported. No formal comparison of the two arms will be conducted. Portions will be reported at 12 months post procedure.
Cardiac Death | 12 Months
  The proportion of patients in each arm that experience Cardiac Death will be summarized and reported. No formal comparison of the two arms will be conducted. Portions will be reported at 12 months post procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Saito, MD, Principal Investigator — Shonan Kamakura General Hospital
Locations (10):
- Japan (10):
  - Iwaki Municipal Iwaki Kyoritsu Hospital, Iwaki, Fukushima
  - Kansai Rosai Hospital, Amagasaki-shi, Hyōgo
  - Tenyokai Central Hospital, Kagoshima, Kagoshima-ken
  - Kanto Rosai Hospital, Kawasaki-shi, Kanagawa
  - Sinkoga Hospital, Kurume-shi, Kurume-shi, Fukuoka
  - Omihachiman Community Medical Center, Ōmihachiman, Shiga
  - Toho Univ.Ohashi Medical Center, Meguro-ku, Tokyo
  - Cardiovascular Institute Hospital, Minato-ku, Tokyo
  - Saiseikai Yokohama Tobu Hospital, Kanagawa, Yokohama
  - Shonan Kamakura General Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: No